CLINICAL TRIAL: NCT05088590
Title: Growing Up Formula Versus Nutritional Supplements: Effect on Catch up Growth, Micronutrient Status, and Solid Foods Intake in Toddlers With Mild or Moderate Malnutrition
Acronym: KEEP Growing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other); Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-3082
Record Dates: First submitted 2021-09-03; First posted 2021-10-22 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Healthy Toddlers 12-36 Months of Age With Mild or Moderate Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growing Up Formula (GUF) (Experimental)
  Interventions: Dietary Supplement: Enfagrow® Neuropro Toddler Nutritional Drink
- Standard Nutritional Supplement (NS) (Active Comparator)
  Interventions: Dietary Supplement: Pediasure® Grow & Gain Protein Shake for Kids

INTERVENTIONS:
Dietary Supplement: Enfagrow® Neuropro Toddler Nutritional Drink — Enfagrow® Neuropro Toddler Nutritional Drink to be consumed per day (equivalent to 40 mL per kg, rounded to the nearest ounce)
  Arms: Growing Up Formula (GUF)
Dietary Supplement: Pediasure® Grow & Gain Protein Shake for Kids — Pediasure® Grow & Gain Protein Shake for Kids to be consumed per day (equivalent to 40 mL per kg, rounded to the nearest ounce)
  Arms: Standard Nutritional Supplement (NS)

SUMMARY:
This is a pilot study to test how a growing-up formula (GUF) compares to a common nutritional supplement (NS), which is regularly used to help toddlers (ages 12-36 months) gain weight. This study will look at whether GUF helps to increase solid food intake for children who are thought to be "picky eaters" and see the effects on growth compared with the NS. To date, it is not clear if GUFs help to increase intake of solid foods. Participants will be placed into one of the two study arms: Enfagrow (GUF) or Pediasure (standard NS).

ELIGIBILITY:
Inclusion Criteria:

Healthy toddlers 12-36 months of age with mild or moderate malnutrition will be defined by at least one of the following indicators:

1. Weight-for-length z-score between -1.0 and -2.9 for children less than 2 years of age using the WHO growth standards; or
2. BMI z-score between -1 to -2.9 for children between 2 and 3 years of age using the CDC growth standards; or
3. Middle upper-arm circumference (MUAC) z-scores between -1 to -2.9 using the WHO growth references; or
4. Percentage of median ideal body weight of 70-89% (using the 50th percentile of the aforementioned growth standards).

Exclusion Criteria:

* Toddlers currently on or with history of tube feeding or with chronic health conditions that influence eating (e.g., food allergies, genetic disorders or developmental disabilities, oral motor difficulties that require sensory or feeding therapy).
* Toddlers who were born at less than 34 weeks gestation, as they may have lingering feeding challenges.
* Toddlers with gastroesophageal reflux disease (GERD) requiring medications or hydrolyzed formula or any type of esophageal disorders will be excluded.
* Toddlers with a history of infant reflux will not be excluded. The PI will make this distinction after a detailed history and record review.
* Families who do not speak English or Spanish in the home.
* Toddlers with suspected malabsorption or conditions that increased metabolic demands such as congenital heart defects.
* Toddlers who have a diagnosed allergy to cow's milk.

The PI will use their clinical discretion to ascertain patient eligibility.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Dietary intake from solid foods - Total proteins in grams | At baseline
  1. Amount of intake of food groups from age-appropriate solid foods;
  2. Intake of calories from age-appropriate solid foods;
  3. Intake of micronutrients from age-appropriate solid foods;
  4. Proportion of calories consumed from age-appropriate solid foods compared with the assigned supplement;
  5. Proportion of micronutrients consumed from age-appropriate solid foods compared with the assigned supplement
Dietary intake from solid foods - Total grains in grams | At baseline
  1. Amount of intake of food groups from age-appropriate solid foods;
  2. Intake of calories from age-appropriate solid foods;
  3. Intake of micronutrients from age-appropriate solid foods;
  4. Proportion of calories consumed from age-appropriate solid foods compared with the assigned supplement;
  5. Proportion of micronutrients consumed from age-appropriate solid foods compared with the assigned supplement
Dietary intake from solid foods - Total vegetables in cups | At baseline
  1. Amount of intake of food groups from age-appropriate solid foods;
  2. Intake of calories from age-appropriate solid foods;
  3. Intake of micronutrients from age-appropriate solid foods;
  4. Proportion of calories consumed from age-appropriate solid foods compared with the assigned supplement;
  5. Proportion of micronutrients consumed from age-appropriate solid foods compared with the assigned supplement
Dietary intake from solid foods - Total proteins in grams | At 3 months
  1. Amount of intake of food groups (total proteins in grams, total grains in grams) from age-appropriate solid foods;
  2. Intake of calories from age-appropriate solid foods;
  3. Intake of micronutrients from age-appropriate solid foods;
  4. Proportion of calories consumed from age-appropriate solid foods compared with the assigned supplement;
  5. Proportion of micronutrients consumed from age-appropriate solid foods compared with the assigned supplement
Dietary intake from solid foods - Total grains in grams | At 3 months
  1. Amount of intake of food groups from age-appropriate solid foods;
  2. Intake of calories from age-appropriate solid foods;
  3. Intake of micronutrients from age-appropriate solid foods;
  4. Proportion of calories consumed from age-appropriate solid foods compared with the assigned supplement;
  5. Proportion of micronutrients consumed from age-appropriate solid foods compared with the assigned supplement
Dietary intake from solid foods - Total vegetables in cups | At 3 months
  1. Amount of intake of food groups from age-appropriate solid foods;
  2. Intake of calories from age-appropriate solid foods;
  3. Intake of micronutrients from age-appropriate solid foods;
  4. Proportion of calories consumed from age-appropriate solid foods compared with the assigned supplement;
  5. Proportion of micronutrients consumed from age-appropriate solid foods compared with the assigned supplement

SECONDARY OUTCOMES:
Secondary Outcomes Measures Related to Growth and Nutrition | Change from baseline to 3 months
  Change in micronutrient status between baseline and month 3 as assessed through circulating micronutrient status, measured by laboratory assessment: CBC, Ferritin, sed rate, zinc, DHA, and vitamin D
Secondary Outcomes Measures Related to Growth and Nutrition -- Weight gain | Change from baseline to 3 months
  Nutrition status assessment - Change in weight Weight gain: catch up growth is defined by weight gain of >6 g per day[

CONTACTS AND LOCATIONS:
Overall Officials: Liliane Diab, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No